CLINICAL TRIAL: NCT05283707
Title: The Effect of "Paula Method Exercises" on the Prevention of Postoperative Distention and Pain Due to Distention After Cesarean Section: A Randomized Controlled Study
Brief Title: The Effect of Paula Method Exercises on Post-cesarean Section Distension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Rabiye DEMIR ISIK, Lecturer, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Akd-3739
Record Dates: First submitted 2022-02-14; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Cesarean Section Complications
Keywords: Distantion; Paula Method Exercises,; Flatulence; Abdominal Pain; Post Cesarean Care; Gas
MeSH Terms: conditions — Flatulence; Abdominal Pain; Mucopolysaccharidosis IV

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): * Continuation of standard post-cesarean section care in the clinic.
  * Implementation of Paula Method Exercises Training Plan 6-8 hours after cesarean section (Paula Method Exercises Practice Card PEUK, Paula Method Exercises Video, Paula Method Exercises Flipcard)
  * Paula Method Exercises; by the researcher, after cesarean section 0.day 6-8 hours, 1st day morning, 2nd day morning.
  * Paula Method Exercises; It was applied by the researcher to the patient on the 0th day 6-8 hours, the 1st day in the morning, and the 2nd day in the morning after the cesarean section.
  * 6-8 hours on day 0, morning on day 1, morning on day 2 after cesarean section Evaluation and recording of bowel sounds before and after Paula Method Exercises, application of "McGill Pain Scale Short Form",
  * Evaluation of first flatulence after cesarean section and first defecation
  Interventions: Behavioral: Paula Method Exercises
- Control Group (No Intervention): * Continuation of standard post-cesarean section care in the clinic.
  * 6-8 hours on day 0, morning on day 1, morning on day 2 after cesarean section Evaluation and recording of bowel sounds, application of "McGill Pain Scale Short Form",
  * Evaluation of first flatulence after cesarean section and first degassing

INTERVENTIONS:
Behavioral: Paula Method Exercises — The Paula Method Exercises were administered by the researcher for 6 to 8 hours, for 10 to 15 minutes on the post-op first day and post-op second day, to women who had a cesarean section.
  Arms: Intervention Group

SUMMARY:
Aim:To examine the effect of "Paula Method Exercises" after cesarean section on the prevention of postoperative distention and pain due to distension.

Method: The study was planned as a double-blind, randomized controlled experimental study.

The study was carried out between November 2021 and February 2022 with women who had undergone cesarean section at Akdeniz University Hospital Gynecology and Obstetrics Clinic and agreed to participate in the study.

The number of individuals to be sampled from the population was determined by the G Power analysis and 80 women were included in the sample.

The data of the study were collected using the Introductory Information Form, the Postoperative Follow-up Form, and the McGill Pain Scale Form.

The women in the intervention group were given training on how to do the Paula Method Exercises in the postoperative period in line with the "Paula Method Exercises Training Plan" by the researcher.

Conclusion: It is predicted that the findings obtained from the data of the study will guide nursing care practices and new researches for the relief of gas and distension after cesarean section.

DETAILED DESCRIPTION:
Aim:To examine the effect of "Paula Method Exercises" after cesarean section on the prevention of postoperative distention and pain due to distension. The gastrointestinal system problems experienced by all individuals undergoing abdominal surgery are important as they affect both the mother and the baby during the post-cesarean section period.

Method: The study was planned as a double-blind, randomized controlled experimental study. The study was carried out between November 2021 and February 2022 with women who had undergone cesarean section at Akdeniz University Hospital Gynecology and Obstetrics Clinic and agreed to participate in the study. The number of individuals to be sampled from the population was determined by the G Power analysis and 80 women were included in the sample. Equal numbers of 80 women who agreed to participate in the study were assigned to the intervention and control groups (https://www.random.org) using the simple randomization method using a simple random numbers table. Women in the intervention and control groups received standard postoperative care in the clinic after cesarean section. In addition, the women in the intervention group were given training on how to do the Paula Method Exercises in the postoperative period in line with the "Paula Method Exercises Training Plan" by the researcher, and the "Paula Method Exercises Card" and "Paula Method Exercises Practice Video" were used, which facilitated the practice of the exercises. Paula Method Exercises were applied to the women in the intervention group by the researcher for 10-15 minutes on postoperative day 0, day 1 and day 2. The data of the study were collected with the "Descriptive Information Form", "Postoperative Follow-up Form" and "McGill Pain Scale Short Form". To both research groups; "Postoperative Follow-up Form" and "McGill Pain Scale Short Form" were applied between 6th and 8th hours, 1st and 2nd days after cesarean section. After the data are collected, the women in the control group will be given Paula Method Exercises training before discharge.

Conclusion: It is predicted that the findings obtained from the data of the study will guide nursing care practices and new researches for the relief of gas and distension after cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-45, who are planned to have an elective Cesarean Section (CD) under spinal anesthesia,
* Admitted to the service within six hours after cesarean section,
* No chronic Charles Bonnet Syndrome (CBS) disease,
* No history of serious (ilostomy, cholastomy, irritable bowel syndrome, etc.) disease related to the gastrointestinal tract,
* Those who volunteered to participate in the study and whose consent was obtained,
* No complications developed during or after the surgery,
* Women who do not have intellectual disability or perception problems and do not have communication difficulties will be included in the study.
* In order not to affect the research results; If there are women in the intervention and control group in the same hospital room, the last woman who was hospitalized in the same room will be excluded from the study.

Exclusion Criteria:

* Enema made,
* Any complication developed and taken to the intensive care unit,
* Not complying with the application process,
* The state of consciousness is not clear / will not be able to participate in the applications,
* Women who cannot communicate for any reason (hearing/speech/hearing, etc.) will be excluded from the research.
* Discharged before two days after cesarean section

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of bowel movements | Bowel sounds will be listened to 6 times. The first measurement will be done between 6-8 hours after cesarean section, the second measurement will be done in the morning on the post-op 1st day, and the third in the morning on the 2nd post-op day.
  An increase in womens' number of bowel movements is a measure of outcome. This increase will be counted by listening with a stethoscope. For the first measurement, bowel sounds will be heard 2 times between 6-8 hours after cesarean section, before and after the intervention. For the second measurement, bowel sounds will be listened to 2 times in the morning on the post-op 1st day after cesarean section, before and after the intervention. For the third measurement, bowel sounds will be listened to 2 times in the morning on the post-op 2nd day after cesarean section, before and after the intervention. Bowel sounds will be listened to 6 times in total. It is predicted that the application of Paula Method Exercises in the postoperative period after cesarean section will decrease the time to pass gas and defecation (in hours) and increase the bowel sounds (in numbers). Significance level is set at p<0.05 in analyzes.
Visual Analogue Scale | Pain will be evaluated 6 times. The first measurement will be made between 6-8 hours after cesarean section, the second measurement will be made in the morning on the 1st postoperative day, and the third in the morning on the 2nd day after the operation.
  Application of Paula Method Exercises in the postoperative period after cesarean section; It is predicted that the Visual Analogue Scale score will decrease in the evaluation of pain due to distention. The minimum value is 0, the maximum value is 10. A low score indicates the success of the attempt. Significance level is set at p<0.05 in analyzes.
First gas extraction time | Until you take your first gas; The first measurement will be made between 6-8 hours after cesarean section, the second will be made on the 1st post-operative day, and the third will be made on the 2nd day after the operation.
  Until the patient has his first gas; The first measurement is between 6-8 hours, the second measurement is made on the 1st day after cesarean section, and the third measurement is made in the morning on the 2nd post-operative day. It is predicted that the application of Paula Method Exercises in the postoperative period after cesarean section will reduce the time of first flatulence. The level of significance in the analyzes was determined as p<0.05.
First defecation extraction time | Until you take your first defecation; The first measurement will be made between 6-8 hours after cesarean section, the second will be made on the 1st post-operative day, and the third will be made on the 2nd day after the operation.
  Until the patient has his first defecation; The first measurement is between 6-8 hours, the second measurement is made on the 1st day after cesarean section, and the third measurement is made in the morning on the 2nd post-operative day. It is predicted that the application of Paula Method Exercises in the postoperative period after cesarean section will reduce the time of first flatulence. The level of significance in the analyzes was determined as p<0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Rabiye Demir Işık, Principal Investigator — Akdeniz Univercity
Locations (1):
- Akdeniz Univercity, Antalya, Konyaaltı, Turkey (Türkiye)

REFERENCES:
- [Background] Liebergall-Wischnitzer M, Hochner-Celnikier D, Lavy Y, Manor O, Shveiky D, Paltiel O. Randomized trial of circular muscle versus pelvic floor training for stress urinary incontinence in women. J Womens Health (Larchmt). 2009 Mar;18(3):377-85. doi: 10.1089/jwh.2008.0950. PMID 19281321
- [Background] Liebergall-Wischnitzer M, Paltiel O, Hochner Celnikier D, Lavy Y, Manor O, Woloski Wruble AC. Sexual function and quality of life of women with stress urinary incontinence: a randomized controlled trial comparing the Paula method (circular muscle exercises) to pelvic floor muscle training (PFMT) exercises. J Sex Med. 2012 Jun;9(6):1613-23. doi: 10.1111/j.1743-6109.2012.02721.x. Epub 2012 Apr 17. PMID 22510279
- [Background] Liebergall-Wischnitzer M, Shvieky D, Lavy Y, Woloski Wruble A, Noble A, Vaknin A. Paula Method (Circular Muscle Exercise) for Urinary Incontinence Symptoms of Women with Multiple Sclerosis: A Pilot Study. J Altern Complement Med. 2020 Jul;26(7):652-653. doi: 10.1089/acm.2020.0069. Epub 2020 May 29. No abstract available. PMID 32471333
- [Background] Liebergall-Wischnitzer M, Shaphir A, Solnica A, Hochner-Celnikier D. Are Paula method exercises effective for gastrointestinal reactivation post-elective cesarean delivery? Randomized controlled trial. J Adv Nurs. 2021 Apr;77(4):2026-2032. doi: 10.1111/jan.14681. Epub 2020 Nov 29. PMID 33249611
- [Background] Liebergall-Wischnitzer M, Hochner-Celnikier D, Lavy Y, Manor O, Arbel R, Paltiel O. Paula method of circular muscle exercises for urinary stress incontinence--a clinical trial. Int Urogynecol J Pelvic Floor Dysfunct. 2005 Sep-Oct;16(5):345-51. doi: 10.1007/s00192-004-1261-6. Epub 2005 Jan 20. PMID 15660184